CLINICAL TRIAL: NCT05847101
Title: Outcome Predictors of Trachea-esophageal Fistula in Neonates Admitted to AUCH
Brief Title: Outcome Predictors of Trachea-esophageal Fistula
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Assem Abd El-razek Elkateeb, Doctor, Assiut University
Other Study IDs: trachea-esophageal fistula
Record Dates: First submitted 2023-04-07; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Tracheo Esophageal Fistula
MeSH Terms: conditions — Tracheoesophageal Fistula

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tracheoesophageal fistula repair — Tracheoesophageal fistula repair

SUMMARY:
In the present study, the investigator aim to evaluate the prevalence, factors affecting outcome and the outcome of neonates with tracheoesophageal fistula.

DETAILED DESCRIPTION:
Tracheoesophageal fistula is a connection between the esophagus and the trachea.

Tracheoesophageal fistula (TEF) represents one of the most common congenital anomalies seen in infants, Infants with TEF classically present with respiratory distress, feeding difficulties, choking, and risk for aspiration. TEF is most commonly associated with other congenital anomalies, particularly cardiac defects. Esophageal atresia (EA) is a related congenital malformation with a similar presentation to TEF and can occur with or without the presence of a fistula.

Although the events leading to separation of the primitive trachea and esophagus are not completely understood, the most commonly accepted hypothesis is that a defect in the lateral septation of the foregut into the trachea and esophagus causes TEF and EA.

The trachea and esophagus develop from a common primitive foregut, and at approximately 4 weeks of gestation, the developing respiratory and gastrointestinal tracts are separated by epithelial ridges. The foregut divides into a ventral respiratory tract and a dorsal esophageal tract; the fistula tract is thought to derive from an embryonic lung bud that fails to undergo branching. These defects of mesenchymal proliferation are thought to lead to TEF formation.

The incidence of TEF is approximately 1 in 3500 births. EA and TEF are classified according to their anatomic configuration.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with tracheoesophageal fistula are/below the age of 28 days.

Exclusion Criteria:

* Patients above the age of 28 days.
* Patients diagnosed with other diseases.
* Patients with acquired tracheoesophageal fistula.

Max Age: 28 Days | Sex: All
Age Groups: Child
Study Population: All newborn admitted to NICU with tracheoesophageal fistula.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Affection of tracheo-esophageal fistula in neanates | Baseline
  evaluate factors affecting outcome of neonates with tracheoesophageal fistula.

REFERENCES:
- [Background] Ma LJ, Xiao Y, Yang QW, Wang J. [Laryngotracheal resection and reconstruction for the treatment of acquired laryngotracheal stenosis]. Zhonghua Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2017 Oct 7;52(10):738-743. doi: 10.3760/cma.j.issn.1673-0860.2017.10.005. Chinese. PMID 29050090
- [Background] Cui PC, Luo JS, Liu Z, Bian K, Guo ZH, Ma RN. [Segmental tracheal resection and anastomosis for the treatment of cicatricial stenosis in cervical tracheal]. Zhonghua Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2016 Feb;51(2):95-9. doi: 10.3760/cma.j.issn.1673-0860.2016.02.004. Chinese. PMID 26898863